CLINICAL TRIAL: NCT02935673
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of Orally Administered Lumicitabine Regimens in Adult Subjects Hospitalized With Respiratory Syncytial Virus
Brief Title: Study to Evaluate the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of Orally Administered Lumicitabine Regimens in Adult Participants Hospitalized With Respiratory Syncytial Virus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108217; 2016-001653-40 (EudraCT Number); 64041575RSV2003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Respiratory Syncytial Viruses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen A (Placebo) (Experimental): Participants of part 1 and part 2 will receive a single loading dose (LD) (Dose 1) followed by 9 maintenance doses (MDs) (Doses 2 to 10) of matching placebo, administered twice daily.
  Interventions: Drug: Placebo
- Regimen B (low-dose lumicitabine) (Experimental): Participants of part 1 and part 2 will receive a single 750 mg LD (Dose 1) followed by nine 250 mg MDs (Doses 2 to 10) of lumicitabine, administered twice daily.
  Interventions: Drug: lumicitabine
- Regimen C (High-dose lumicitabine) (Experimental): Participants of part 2 will receive a single 1000 mg LD (Dose 1) followed by nine 500 mg MDs (Doses 2 to 10) of lumicitabine, administered twice daily.
  Interventions: Drug: lumicitabine

INTERVENTIONS:
Drug: lumicitabine — Oral administration of lumicitabine as tablet.
  Other Names: ALS-8176/JNJ-64041575
  Arms: Regimen B (low-dose lumicitabine); Regimen C (High-dose lumicitabine)
Drug: Placebo — Oral administration of matching placebo.
  Arms: Regimen A (Placebo)

SUMMARY:
The purpose of this study is to characterize the Pharmacokinetic and to confirm the popPK model derived from healthy volunteers in hospitalized adults who are infected with respiratory syncytial virus (RSV) and to determine in adults who are hospitalized with respiratory syncytial virus (RSV) infection the dose response relationship of multiple regimens of lumicitabine on antiviral activity based on nasal RSV shedding using quantitative real-time reverse transcriptase-polymerase chain reaction (qRT-PCR) assay.

DETAILED DESCRIPTION:
The study will be conducted in 3 phases: a screening phase, a treatment phase from Day 1 to Day 5/6 (depending on the timing of the loading dose), and a follow-up phase for a total of 28 days post randomization. Participants will have assessments completed at Day 7, Day 10, Day 14, and Day 28. Depending on discharge date, assessments will be completed either while hospitalized or during outpatient visits. The duration of the participant's participation will be approximately 28 days. The study will be performed in 2 parts. Participants will be randomly assigned to one of 2 treatment groups in part 1, and to one of 3 treatment groups in part 2. Treatment groups will be evaluated for PK and safety after a target of approximately 24 participants have been enrolled in part 1 and before initiating part 2 (approximately 90 participants in part 2). An Independent Data Monitoring Committee (IDMC) will be established to monitor the safety of participants and will review data in an unblinded manner on a regular basis to ensure the continuing safety of the participants enrolled in this study and to evaluate whether efficacy objectives are met. The committee will meet periodically to review interim data. Based on the recommendations of the IDMC following interim analyses/reviews, an increase in duration may be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized (or in emergency room prior to hospitalization) at the time of randomization and unlikely to be discharged for the first 24 hours after randomization
* Diagnosed with respiratory syncytial virus (RSV) infection based on polymerase chain reaction (PCR)-based assay with or without co infection with another respiratory pathogen (eg, influenza, human metapneumovirus, or bacteria)
* With the exception of the RSV disease, medically stable on the basis of medical history, physical examination, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population and/or the RSV infection. This determination must be recorded in the participant's source documents and initialed by the investigator
* A woman must have a negative urine beta human chorionic gonadotropin at screening
* A woman must agree not to donate eggs (ova, oocytes) during the study and for at least 44 days after receiving the last dose of study drug
* Contraceptive use by women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies A woman must be of non-childbearing potential defined as either: a) Postmenopausal: a postmenopausal state is defined as more than (>) 45 years and no menses for 12 consecutive months without an alternative medical cause, OR Permanently sterile: permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures (without reversal operation), and bilateral oophorectomy. b) Of childbearing potential and, if heterosexually active, also included: practicing a highly effective method of contraception (failure rate of less than (<) 1percent (%) per year when used consistently and correctly)
* Participants must have a body weight of at least 50.0 kilogram, at screening

Exclusion Criteria:

* Participants who are not expected to survive for more than 48 hours
* Participants who have had major thoracic or abdominal surgery in the 6 weeks prior to randomization
* Participants who are considered by the investigator to be immuno-compromised within the past 12 months, whether due to underlying medical condition (example, malignancy or genetic disorder) or medical therapy (example, medications other than corticosteroids for the treatment of chronic obstructive pulmonary disease (COPD) or asthma exacerbations, chemotherapy, radiation, stem cell or solid organ transplant)
* Participants with a known history of human immunodeficiency virus (HIV) or chronic viral hepatitis
* Participants undergoing peritoneal dialysis, hemodialysis, or hemofiltration or with an estimated glomerular filtration rate (GFR, determined by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) of (<) 60 milliliters per minute (mL/min) per 1.73 meter square (m^2)
* Participants with 1 or more of the following laboratory abnormalities at screening as defined by the Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table: Hemoglobin <9.5 gram per deciliter (g/dL), Platelet count <75,000 per millimeter cube (/mm^³), White blood cell count <1,000/mm^³, Absolute neutrophil count <1,000/mm^³

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (109):
- United States (10):
  - Fresno, California
  - Orange, California
  - Stanford, California
  - Eustis, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - St Louis, Missouri
  - Butte, Montana
  - Rochester, New York
  - Syracuse, New York
- Argentina (8):
  - Bahía Blanca
  - Barrio Parque Velez Sarfield
  - Buenos Aires
  - Ciudad de Buenos Aires
  - Ciudad de La Plata
  - Córdoba
  - La Plata
  - Rosario
- Australia (5):
  - Cairns
  - Geelong
  - Melbourne
  - South Brisbane
  - Sydney
- Belgium (2):
  - Bruges
  - Lier
- Brazil (5):
  - Belo Horizonte
  - Passo Fundo
  - Porto Alegre
  - Ribeirão Preto
  - São Paulo
- Bulgaria (5):
  - Kozloduy
  - Petrich
  - Rousse
  - Sofia
  - Veliko Tarnovo
- Canada (2):
  - Hamilton, Ontario
  - Toronto, Ontario
- France (11):
  - Colombes
  - Dijon
  - La Tronche
  - Limoges
  - Lyon
  - Morlaix
  - Nantes
  - Paris
  - Poitiers
  - Suresnes
  - Tours
- Germany (2):
  - Marburg
  - Witten
- Japan (21):
  - Fukuoka
  - Fukushima
  - Funaishikawa
  - Gifu
  - Gunma
  - Hamamatue
  - Isahaya
  - Izumo
  - Kitakyushu
  - Kobe
  - Nagasaki
  - Nagoya
  - Osaka
  - Ōta-ku
  - Sendai
  - Seto
  - Shiogama
  - Tanabe
  - Tokyo
  - Tsu
  - Uruma
- Malaysia (7):
  - Johor Bharu
  - Kuala
  - Kuala Lumpur
  - Kuching
  - Malacca
  - Miri
  - Taiping
- Mexico (4):
  - Cuernavaca
  - Guadalajara
  - México
  - Monterrey
- Netherlands (2):
  - Leiden
  - Utrecht
- Poland (4):
  - Bialystok
  - Chęciny
  - Mrozy
  - Proszowice
- South Korea (6):
  - Bucheon-si
  - Daegu
  - Gwangju
  - Incheon
  - Seongnam
  - Seoul
- Spain (5):
  - Elche
  - Granada
  - Madrid
  - Santiago de Compostela
  - Vigo
- Sweden (4):
  - Gothenburg
  - Malmo
  - Umeå
  - Uppsala
- Taiwan (4):
  - Kaohsiung City
  - New Taipei City
  - Tainan
  - Taipei
- United Kingdom (2):
  - London
  - Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sponsor halted screening and enrollment in study on 22 June 2018 due to emerging lumicitabine nonclinical data. On 17 October 2018, study was stopped prematurely by sponsor as a precautionary measure, to allow further evaluation of new nonclinical pharmacokinetic (PK) and safety findings and determine their relevance to human studies.
Pre-assignment Details: A total of 49 participants were randomized and treated (2 participants in Part 0, 36 participants in Part 1 and 11 participants in Part 2). Analyses were conducted on pooled groups across the 3 study parts.
Groups:
- Placebo: Participants received a single loading dose (LD) (Dose 1) of matching placebo tablet orally on Day 1 followed by nine maintenance doses (MD) (Doses 2 to 10) of matching placebo tablets orally twice daily (bid) from Day 1/2 to Day 5/6 (depending on the timing of the LD administration).
- 750 mg LD / 250 mg MD Lumicitabine: Participants received a single 750 milligram (mg) LD (Dose 1) of lumicitabine tablet orally followed by nine MD (Doses 2 to 10) of 250 mg lumicitabine tablets orally bid from Day 1/2 to Day 5/6 (depending on the timing of the LD administration).
- 1000 mg LD / 500 mg MD Lumicitabine: Participants received a single 1000 mg LD (Dose 1) of lumicitabine tablet orally followed by nine MD (Doses 2 to 10) of 500 mg lumicitabine tablets orally bid from Day 1/2 to Day 5/6 (depending on the timing of the LD administration).
Period: Overall Study
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Started | 16 | 27 | 6
Completed | 15 | 24 | 6
Not Completed | 1 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine | Total
Number analyzed (Participants) | 16 | 27 | 6 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (17.94) | 66.3 (17.75) | 68.7 (18.46) | 66.3 (17.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 5 | 19
  Male | 11 | 18 | 1 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 14 | 25 | 6 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 11 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 14 | 3 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 2 | 0 | 0 | 2
  AUSTRALIA | 3 | 3 | 1 | 7
  FRANCE | 1 | 6 | 0 | 7
  JAPAN | 3 | 3 | 3 | 9
  MALAYSIA | 0 | 2 | 0 | 2
  POLAND | 0 | 2 | 0 | 2
  SOUTH KOREA | 1 | 3 | 0 | 4
  SPAIN | 1 | 2 | 0 | 3
  SWEDEN | 3 | 2 | 2 | 7
  TAIWAN | 0 | 3 | 0 | 3
  UNITED KINGDOM | 1 | 0 | 0 | 1
  UNITED STATES | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of JNJ-63549109 at Day 1
Description: Cmax is the maximum observed plasma concentration of JNJ-63549109. JNJ-63549109 is the metabolized product of lumicitabine.
Time Frame: Day 1
Population: Pharmacokinetic (PK) analysis was performed on safety set which included all participants who received at least 1 dose of study drug, analyzed as treated. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 26 | 4
nanogram per milliliter (ng/mL) | 1845 (545.2) | 2801 (1509)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of JNJ-63549109 at Day 5
Description: as for outcome 1
Time Frame: Day 5
Population: PK analysis was performed on safety set which included all participants who received at least 1 dose of study drug, analyzed as treated. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 22 | 2
ng/mL | 745.4 (164.2) | 1145 (440.8)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours After Dosing (AUC[0-24h]) of JNJ-63549109 at Day 1
Description: AUC(0-24) is the area under the plasma concentration-time curve from time 0 to 24 hours after dosing of JNJ-63549109. JNJ-63549109 is the metabolized product of lumicitabine.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 26 | 4
nanogram*hour per milliliter (ng*h/mL) | 9936 (2090) | 17120 (4330)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours After Dosing (AUC[0-24h]) of JNJ-63549109 at Day 5
Description: as for outcome 3
Time Frame: Day 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 22 | 2
ng*h/mL | 7557 (1525) | 13300 (4603)

5. Primary Outcome: Trough Observed Plasma Concentration (Ctrough) of JNJ-63549109 at Day 1
Description: Ctrough is the trough observed plasma concentration of JNJ-63549109. JNJ-63549109 is the metabolized product of lumicitabine.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 26 | 4
ng/mL | 93.7 (44.16) | 184.4 (70.66)

6. Primary Outcome: Trough Observed Plasma Concentration (Ctrough) of JNJ-63549109 at Day 5
Description: as for outcome 5
Time Frame: Day 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 22 | 2
ng/mL | 148.3 (60.41) | 281.3 (156.6)

7. Primary Outcome: Least Square Mean Difference (Low and High Dose Lumicitabine Versus Placebo) of Respiratory Syncytial Virus (RSV) Ribonucleic Acid (RNA) Viral Load Area Under the Concentration-time Curve From Day 1 to 7 (AUC[1-7])
Description: RSV RNA viral load in log10 copies/milliliter/day (log10 copies/mL/day) was measured in mid-turbinate nasal swabs and in endotracheal samples (obtained from intubated participants or via suction through tracheostomy or other sampling methods) using quantitative reverse transcription-polymerase chain reaction (qRT-PCR). Due to early termination of study, the analysis was not conducted as planned. Instead, using the same specification as for the primary analysis, a comparison was made on the AUC(1-7) days of pooled active treatment groups versus pooled placebo. The comparison was done as planned using a mixed model for repeated measures, using all available viral load data of baseline up to and including Day 7. The model computes the AUC at group level based on all available data, taking missing data into account under the missing at random assumption. The table reports the planned difference versus (pooled) placebo. No adjustment for multiplicity was applied.
Time Frame: Day 1 (Baseline) to 7
Population: Intent-to-treat-infected (ITT-i) set included all randomly assigned participants who received at least 1 dose of study drug and who had an RSV infection confirmed by a PCR-based assay at the central laboratory at baseline, analyzed as randomized. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL/day
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
log10 copies/mL/day
  Day 2 | -0.3 [-0.9 to 0.3] | -1.4 [-2.0 to -0.9] | -2.5 [-3.6 to -1.3]
  Day 3 | -1.4 [-2.1 to -0.7] | -1.9 [-2.5 to -1.2] | -1.9 [-3.4 to -0.5]
  Day 4 | -2.1 [-2.8 to -1.4] | -2.2 [-2.8 to -1.6] | -1.8 [-3.2 to -0.5]
  Day 5 | -2.5 [-3.2 to -1.9] | -2.5 [-3.1 to -1.9] | -1.3 [-2.6 to -0.1]
  Day 6 | -2.5 [-3.2 to -1.7] | -2.7 [-3.3 to -2.0] | -3.1 [-4.5 to -1.7]
  Day 7 | -2.8 [-3.5 to -2.0] | -2.8 [-3.5 to -2.2] | -3.3 [-4.5 to -2.0]
Statistical Analysis 1: Comparison: Placebo vs 750 mg LD / 250 mg MD Lumicitabine; Test type: Superiority; AUC(1-7) difference vs (pooled) placebo = -0.32, 95% CI 2-sided [-0.89 to 0.24]; Mixed model for repeated measures, using all available viral load data of baseline and up to and including Day 7, taking missing data into account under the missing at random assumption
Statistical Analysis 2: Comparison: Placebo vs 1000 mg LD / 500 mg MD Lumicitabine; Test type: Superiority; AUC(1-7) difference vs (pooled) placebo = -0.36, 95% CI 2-sided [-1.33 to 0.62]; [other analysis details as in outcome 7, analysis 1]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Time Frame: Up to 28 Days
Population: Safety set included all participants who received at least 1 dose of study drug, analyzed as treated. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 16 | 27 | 6
Participants | 7 | 22 | 5

9. Secondary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Number of participants with vital sign (systolic and diastolic blood pressure [BP], pulse rate, respiratory rate, temperature and oxygen saturation) abnormalities were reported. For systolic BP: abnormally low refers to less than or equal to (<=) 90 millimeter of mercury (mmHg); for diastolic BP: abnormally low refers to <= 50 mmHg; for pulse rate abnormally low refers to less than (<) 45 beats per minutes (bpm) and abnormally high refers to greater than or equal to (>=) 120 bpm; for temperature in degree Celsius abnormally high refers to greater than (>) 37.8 (tympanic), >38.0 (forehead), >38.0 (oral), >37.2 (rectal), >38.0 (axillary); for oxygen saturation in percentage (%) abnormally low refers to < 95. Grade 1 = mild; grade 2 = moderate; grade 3 = severe.
Time Frame: Up to 28 Days
Population: Safety set included all participants who received at least 1 dose of study drug, analyzed as treated. Here 'n' (number analyzed) signifies number of participants evaluable for specified categories. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 16 | 27 | 6
Participants
  Systolic BP (Abnormally low) | 1 | 0 | 0
  Systolic BP (Grade 1 or mild) | 2 | 6 | 2
  Systolic BP (Grade 2 or moderate) | 5 | 4 | 0
  Systolic BP (Grade 3 or severe) | 1 | 1 | 1
  Diastolic BP (Abnormally low) | 2 | 1 | 1
  Diastolic BP (Grade 1 or mild) | 5 | 8 | 1
  Diastolic BP (Grade 2 or moderate) | 3 | 1 | 0
  Diastolic BP (Grade 3 or severe) | 0 | 1 | 0
  Pulse Rate (Abnormally high) | 2 | 1 | 0
  Respiratory Rate (Grade 1 or mild): number analyzed (Participants) | 16 | 26 | 6
  Respiratory Rate (Grade 1 or mild) | 2 | 0 | 1
  Respiratory Rate (Grade 2 or moderate): number analyzed (Participants) | 16 | 26 | 6
  Respiratory Rate (Grade 2 or moderate) | 4 | 6 | 1
  Respiratory Rate (Grade 3 or severe): number analyzed (Participants) | 16 | 26 | 6
  Respiratory Rate (Grade 3 or severe) | 3 | 2 | 0
  Temperature (Abnormally high) | 4 | 2 | 0
  Oxygen Saturation (Abnormally low) | 7 | 9 | 2

10. Secondary Outcome: Number of Participants With QT Interval Abnormalities
Description: Number of participants with QT interval abnormalities (prolonged) were reported.
Time Frame: Up to 28 Days
Population: Safety set included all participants who received at least 1 dose of study drug, analyzed as treated. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 24 | 5
Participants | 0 | 1 | 0

11. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Number of participants with clinical laboratory (serum chemistry and hematology) abnormalities were reported. Abbreviations; Erythrocyte MCHC = Erythrocyte Mean Corpuscular Hemoglobin Concentration; Erythrocyte MCH = Erythrocyte Mean Corpuscular Hemoglobin; Ery. = Erythrocyte
Time Frame: Up to 28 Days
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 16 | 27 | 6
Participants
  Bicarbonate : Low: number analyzed (Participants) | 9 | 17 | 2
  Bicarbonate : Low | 0 | 2 | 0
  Bicarbonate: High: number analyzed (Participants) | 9 | 17 | 2
  Bicarbonate: High | 3 | 5 | 0
  Chloride : Low: number analyzed (Participants) | 15 | 25 | 6
  Chloride : Low | 0 | 3 | 0
  Chloride : High: number analyzed (Participants) | 15 | 25 | 6
  Chloride : High | 0 | 2 | 0
  Creatine Kinase : Low: number analyzed (Participants) | 13 | 19 | 6
  Creatine Kinase : Low | 4 | 2 | 3
  Creatine Kinase ; High: number analyzed (Participants) | 13 | 19 | 6
  Creatine Kinase ; High | 0 | 0 | 1
  Direct Bilirubin : High: number analyzed (Participants) | 7 | 15 | 4
  Direct Bilirubin : High | 0 | 1 | 0
  Indirect Bilirubin : Low: number analyzed (Participants) | 7 | 12 | 4
  Indirect Bilirubin : Low | 1 | 0 | 2
  Basophils : High | 0 | 0 | 1
  Eosinophils : High | 3 | 1 | 1
  Erythrocytes MCHC : Low | 1 | 1 | 0
  Erythrocytes MCH : Low | 1 | 0 | 0
  Erythrocytes MCH : High | 0 | 3 | 1
  Erythrocytes : Low | 5 | 3 | 1
  Ery. Distribution Width : Low: number analyzed (Participants) | 11 | 20 | 4
  Ery. Distribution Width : Low | 0 | 1 | 0
  Ery. Distribution Width : High: number analyzed (Participants) | 11 | 20 | 4
  Ery. Distribution Width : High | 2 | 5 | 3
  Hematocrit : Low: number analyzed (Participants) | 16 | 26 | 6
  Hematocrit : Low | 4 | 5 | 0
  Hematocrit : High: number analyzed (Participants) | 16 | 26 | 6
  Hematocrit : High | 1 | 0 | 0
  Lymphocytes : Low | 0 | 4 | 0
  Lymphocytes : High | 4 | 3 | 2
  Monocyte : Low | 0 | 2 | 1
  Monocyte : High | 5 | 5 | 3
  Reticulocytes : Low: number analyzed (Participants) | 8 | 11 | 6
  Reticulocytes : Low | 0 | 1 | 2
  Reticulocytes : High: number analyzed (Participants) | 8 | 11 | 6
  Reticulocytes : High | 4 | 2 | 4
  Reticulocytes/Erythrocytes : Low: number analyzed (Participants) | 6 | 14 | 4
  Reticulocytes/Erythrocytes : Low | 1 | 0 | 1
  Reticulocytes/Erythrocytes : High: number analyzed (Participants) | 6 | 14 | 4
  Reticulocytes/Erythrocytes : High | 4 | 9 | 3

12. Secondary Outcome: Time of Hospital Stay From Study Treatment Initiation to Discharge
Description: It is the time from treatment initiation to hospital discharge in hours.
Time Frame: From study treatment initiation to discharge (Up to 28 Days)
Population: ITT-i set included all randomly assigned participants who received at least 1 dose of study drug and who had an RSV infection confirmed by a PCR-based assay at the central laboratory at baseline, analyzed as randomized. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Hours | 183.91 (217.020) | 146.72 (94.910) | 405.24 (294.771)

13. Secondary Outcome: Time of Hospital Stay From Admission to Discharge
Description: It is the time from hospital admission to hospital discharge in hours.
Time Frame: From admission to discharge (Up to 28 Days)
Population: Analysis was performed on ITT-i set. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 10 | 17 | 3
Hours | 192.40 (199.363) | 181.97 (107.938) | 297.53 (348.729)

14. Secondary Outcome: Time of Hospital Stay From Study Treatment Initiation to Readiness for Discharge
Description: It is the time from study treatment initiation to readiness for discharge in hours, with readiness for discharge defined by the investigator.
Time Frame: From study treatment initiation to readiness for discharge on Day 2 or up to Day 6 if hospitalization is prolonged
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Hours | 111.05 (78.237) | 144.17 (96.019) | 197.60 (256.702)

15. Secondary Outcome: Time of Hospital Stay From Admission to Readiness for Discharge
Description: It is the time from hospital admission to readiness for discharge in hours, with readiness for discharge defined by the investigator.
Time Frame: Up to 28 Days
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 10 | 17 | 3
Hours | 133.41 (83.057) | 178.82 (108.522) | 297.13 (349.159)

16. Secondary Outcome: Number of Participants Who Required to be Admitted to the Intensive Care Unit (ICU) Since Initiation of Treatment
Description: Number of participants who required to be admitted to the ICU since initiation of treatment were reported.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Participants | 0 | 0 | 0

17. Secondary Outcome: Duration of Intensive Care Unit Stay
Description: In the event that a participant required ICU since initiation of treatment, the duration for how long the participant remained in the ICU was measured.
Time Frame: Up to 28 Days
Population: ITT-i set included all randomly assigned participants who received at least 1 dose of study drug and who had an RSV infection confirmed by a PCR-based assay at the central laboratory at baseline, analyzed as randomized. Overall number of participants analyzed is 0, since none of the participants were admitted to ICU since initiation of treatment.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Number of Participants Who Required Supplemental Oxygen
Description: Number of participants who required supplemental oxygen were reported.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Participants | 14 | 18 | 4

19. Secondary Outcome: Time to End of Oxygen Supplementation
Description: It is the time from first dose of study drug to the last end date and time of any oxygen supplementation in hours.
Time Frame: Up to 28 Days
Population: Population included ITT-i set who required supplemental oxygen. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 14 | 18 | 4
Hours | 83.92 (168.125) | 139.38 (237.584) | 132.40 (288.568)

20. Secondary Outcome: Time (Number of Hours) Until Peripheral Capillary Oxygen Saturation (SpO2) Greater Than or Equal to (>=) 93 Percent (%) on Room Air Among Participants Who Were Not on Supplemental Oxygen Prior to the Onset of Respiratory Symptoms
Description: Time (number of hours) until SpO2 >= 93% on room air among participants who were not on supplemental oxygen prior to the onset of respiratory symptoms was reported.
Time Frame: Up to 28 Days
Population: Data was not collected and analyzed because this study was stopped prematurely.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Time to Return to Pre-respiratory Syncytial Virus (Pre-RSV) Disease Level for Respiratory Rate
Description: It is the time from first dose of study drug until the time to return to pre-RSV disease level for respiratory rate. The return to pre-RSV disease level occurred when the observed value of the parameter was indicated by the investigator as normal, and no later observed values were indicated by the investigator as abnormal.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Hours | 64.72 (180.542) | 47.75 (153.293) | 196.96 (290.694)

22. Secondary Outcome: Time to Return to Pre-RSV Disease Level for Oxygen Saturation
Description: It is the time from first dose of study drug until the time to return to pre-RSV disease level for oxygen saturation. The return to pre-RSV disease level occurred when the observed value of the parameter was indicated by the investigator as normal, and no later observed values were indicated by the investigator as abnormal.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Hours | 55.55 (85.915) | 33.85 (57.703) | 47.56 (106.347)

23. Secondary Outcome: Time to Return to Pre-RSV Disease Level for Body Temperature
Description: It is the time from first dose of study drug until the time to return to pre-RSV disease level for body temperature. The return to pre-RSV disease level occurred when the observed value of the parameter was indicated by the investigator as normal, and no later observed values were indicated by the investigator as abnormal.
Time Frame: Up to 28 Days
Population: Data was not collected and analyzed because this study was stopped prematurely.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Number of Participants Who Required Noninvasive Mechanical Ventilation Support
Description: Number of participants who required noninvasive mechanical ventilation support (that is supplemental oxygen [excluding mechanical ventilation]) were reported.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Participants | 14 | 18 | 4

25. Secondary Outcome: Time to End of Noninvasive Mechanical Ventilation Support
Description: It is the time from first dose of study drug to the last end date and time of noninvasive mechanical ventilation support in hours.
Time Frame: Up to 28 Days
Population: Population included ITT-i set who required noninvasive mechanical ventilation support. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 14 | 18 | 4
Hours | 83.92 (168.125) | 139.38 (237.584) | 132.40 (288.568)

26. Secondary Outcome: Number of Participants Who Required Invasive Mechanical Ventilation Support
Description: Number of participants who required invasive mechanical ventilation support were reported.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Participants | 0 | 0 | 0

27. Secondary Outcome: Time to End of Invasive Mechanical Ventilation Support
Description: It is the time from first dose of study drug to the last end date and time of invasive mechanical ventilation support in hours.
Time Frame: Up to 28 Days
Population: ITT-i set included all randomly assigned participants who received at least 1 dose of study drug and who had an RSV infection confirmed by a PCR-based assay at the central laboratory at baseline, analyzed as randomized. Overall number of participants analyzed is zero, since none of the participants required mechanical ventilation support.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Time to Return to Pre-RSV Functional Status as Assessed by KATZ Activities of Daily Living (ADL) Score
Description: It is the time from first dose of study drug until the time to return to pre-RSV functional status. Functional status is the total points on the KATZ index of independence in activities of daily living (KATZ ADL score). Katz activities of daily living assessed questions related to bathing, dressing, toileting, transferring, continence and feeding components. Total score was calculated by adding the scores for all 6 activities which ranges from 0 high (participant independent) to 6 low (participant very dependent). If one or more component was missing, then the KATZ ADL score was not calculated. The return to pre-RSV functional status occurs at the timepoint where for the first time the KATZ ADL score is equal or higher than the pre-RSV KATZ ADL score and after which no scores lower than the pre-RSV KATZ ADL score occur anymore.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Days | 3.60 (7.434) | 4.48 (6.961) | 6.00 (11.203)

29. Secondary Outcome: Number of Participants Who Required Hydration or Feeding by Intravenous (IV) Catheter or Nasogastric Tube
Description: Number of participants who required hydration or feeding by IV catheter or nasogastric tube were reported.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Participants | 3 | 5 | 1

30. Secondary Outcome: Time to Clinical Stability
Description: Time to clinical stability is defined as the time from first dose of study drug until the time at which the following criteria were all met: normalization of blood oxygen level (return to baseline; by pulse oximetry) without requirement of supplemental oxygen beyond baseline level, normalization of oral feeding, normalization of respiratory rate and normalization of heart rate.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Hours | 151.21 (266.460) | 171.74 (261.384) | 207.00 (282.955)

31. Secondary Outcome: Number of Participants in Each Ordinal Scale Category
Description: Number of participants in each ordinal scale category were reported. Ordinal scale consists of 6 categories or clinical states that are exhaustive, mutually exclusive, and ordered: category 1) death; category 2) admitted to ICU; category 3) non-ICU hospitalization requiring supplemental oxygen; category 4) non-ICU hospitalization not requiring supplemental oxygen; category 5) not hospitalized, unable to resume normal activities; category 6) not hospitalized, resumption of normal activities.
Time Frame: Day 5/6 (Day of last study treatment)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Participants
  Category 1 | 0 | 0 | 0
  Category 2 | 0 | 1 | 0
  Category 3 | 2 | 5 | 1
  Category 4 | 6 | 8 | 1
  Category 5 | 5 | 2 | 1
  Category 6 | 2 | 5 | 2

32. Secondary Outcome: Number of Participants With All-Cause Mortality
Description: All-cause mortality included all deaths of participants due to any cause.
Time Frame: Up to 28 Days
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 16 | 27 | 6
Participants | 0 | 0 | 0

33. Secondary Outcome: RSV RNA Viral Load Over Time
Description: Antiviral activity RSV RNA viral load was measured in mid-turbinate nasal swabs (obtained from non-intubated participants) or in mid-turbinate nasal swabs and endotracheal samples (obtained from intubated participants or via suction through tracheostomy or other sampling methods) using qRT-PCR performed at the central laboratory.
Time Frame: Days 2, 3, 4, 5, 6, 7, 10, 14, and 28
Population: Analysis was performed on ITT-i set. Here 'n' (number analyzed) signifies number of participants evaluable for each time point. Analyses were conducted on pooled groups across the 3 study parts.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
log10 copies/mL
  Day 2: number analyzed (Participants) | 15 | 21 | 4
  Day 2 | 5.9257 (1.95951) | 4.7208 (1.60154) | 3.4242 (1.10867)
  Day 3: number analyzed (Participants) | 15 | 19 | 3
  Day 3 | 4.8255 (1.84651) | 4.3515 (1.97633) | 4.3129 (0.99078)
  Day 4: number analyzed (Participants) | 15 | 21 | 3
  Day 4 | 4.0608 (1.57493) | 3.9345 (1.64600) | 4.0729 (1.15419)
  Day 5: number analyzed (Participants) | 15 | 20 | 3
  Day 5 | 3.6463 (1.44056) | 3.6206 (1.71515) | 4.5344 (0.97473)
  Day 6: number analyzed (Participants) | 15 | 19 | 3
  Day 6 | 3.6996 (1.98383) | 3.4313 (1.57700) | 3.2163 (1.30083)
  Day 7: number analyzed (Participants) | 15 | 19 | 5
  Day 7 | 3.4044 (1.75773) | 3.2306 (1.58432) | 2.6147 (0.89779)
  Day 10: number analyzed (Participants) | 15 | 15 | 4
  Day 10 | 2.5966 (1.04644) | 2.7516 (1.72825) | 2.5792 (1.00954)
  Day 14: number analyzed (Participants) | 15 | 21 | 4
  Day 14 | 2.3605 (1.00220) | 2.3010 (1.03732) | 2.1512 (0.50236)
  Day 28: number analyzed (Participants) | 14 | 21 | 4
  Day 28 | 1.9179 (0.06682) | 1.9714 (0.22559) | 1.9000 (0.00000)

34. Secondary Outcome: Peak Viral Load
Description: Peak Viral load is the highest value of log10 viral load at or after the baseline measurement. Peak viral load over time was measured by qRT-PCR.
Time Frame: Up to 28 Days
Population: Data was not collected and analyzed because this study was stopped prematurely.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: Time to Peak Viral Load
Description: Time to peak viral load is the time from initiation of study treatment until the first time point with the peak viral load.
Time Frame: Up to 28 Days
Population: Data was not collected and analyzed because this study was stopped prematurely.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

36. Secondary Outcome: Rate of Decline of Viral Load
Description: Rate of decline of viral load over the first 24 hours calculated as a log decline/24 hours defined as: 24-hour log viral load after first dose of study drug minus (-) log viral load at baseline divided by (/) date/time of 24-hour viral load sample - date/time of baseline viral load.
Time Frame: Up to 28 Days
Population: Data was not collected and analyzed because this study was stopped prematurely.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

37. Secondary Outcome: Time to RSV RNA Viral Load Being Undetectable
Description: It is the time in hours from initiation of study treatment until the first post baseline time point at which the virus is undetectable in an assessment and after which time no detectable virus assessment follows as measured by qRT-PCR.
Time Frame: Up to 28 Days
Population: Data was not collected and analyzed because this study was stopped prematurely.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

38. Secondary Outcome: Number of Participants With Undetectable Viral Load
Description: Number of participants with undetectable viral load up to 28 days were reported.
Time Frame: Up to 28 Days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 15 | 21 | 5
Participants | 14 | 19 | 5

39. Secondary Outcome: RSV RNA Viral Load AUC up to Day 14
Description: RSV RNA viral load was measured in midturbinate nasal swabs and in endotracheal samples (obtained from intubated participants or via suction through tracheostomy or other sampling.
Time Frame: Up to Day 14
Population: Data was not collected and analyzed because this study was stopped prematurely.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

40. Secondary Outcome: RSV RNA Viral Load AUC in Participants Assigned to a Longer Dosing Duration
Description: as for outcome 39
Time Frame: Up to 1 Day after the last dose of study drug
Population: ITT-i set included all randomly assigned participants who received at least 1 dose of study drug and who had an RSV infection confirmed by a PCR-based assay at the central laboratory at baseline, analyzed as randomized. No participant received extended treatment, therefore data was not analyzed.
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 0 | 0 | 0

41. Secondary Outcome: Number of Participants With Postbaseline Changes in the RSV Polymerase L Gene and Other Regions of the RSV Genome Compared With Baseline Sequences
Description: Number of participants with postbaseline changes in the RSV polymerase L gene and other regions of the RSV genome compared with baseline sequences were reported.
Time Frame: Baseline up to 28 Days
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
Number analyzed (Participants) | 10 | 12 | 4
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 Days
Arm/Group | Placebo | 750 mg LD / 250 mg MD Lumicitabine | 1000 mg LD / 500 mg MD Lumicitabine
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/27 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/16 | 4/27 | 1/6
Other Adverse Events (participants affected / at risk) | 6/16 | 17/27 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | 750 mg LD / 250 mg MD Lumicitabine (N=27) | 1000 mg LD / 500 mg MD Lumicitabine (N=6)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | 750 mg LD / 250 mg MD Lumicitabine (N=27) | 1000 mg LD / 500 mg MD Lumicitabine (N=6)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 2 | 2 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 2 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection Bacterial (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 3 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 2 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 2 | 0
Blood Fibrinogen Increased (Investigations) | 1 | 0 | 0
C-Reactive Protein Increased (Investigations) | 1 | 0 | 0
Eosinophil Count Increased (Investigations) | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 1 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1
Occult Blood Positive (Investigations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
As the study was stopped prematurely the planned final analyses were adapted. Due to small number of participants in Part 2, it was decided to pool the data from the 3 parts of the study to perform an evaluation of selected planned analyses only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT02935673/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT02935673/SAP_001.pdf